CLINICAL TRIAL: NCT00605943
Title: Pilot Study for the Detection of Neutralizing Antibodies in Patients Treated With Bevacizumab Avastin or Ranibizumab Lucentis
Brief Title: Detection of Neutralizing Antibodies in Patients Treated With Bevacizumab or Ranibizumab
Status: Completed | Type: Observational
Sponsor: National Eye Institute (NEI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 080061; 08-EI-0061
Record Dates: First submitted 2008-01-23; First posted 2008-01-31 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2009-08-04

CONDITIONS: Macular Degeneration
Keywords: Retinal Disease; Bevacizumab; Ranibizumab; Retinal Eye Disease; Macular Degeneration
MeSH Terms: conditions — Macular Degeneration; Retinal Diseases

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
This study will measure antibody levels in the blood of people with bleeding or swelling in the retina who have or have not been treated with bevacizumab (Avastin[Trademark]or ranibizumab (Lucentis[Trademark]). These drugs have been useful in reducing retinal bleeding and swelling in people with eye diseases that cause these symptoms, but the drugs' effects usually wear off and they have to be given repeatedly. In some patients, the benefits become less and less. It is possible that over time, patients taking these drugs may produce antibodies that act against the drugs, thus neutralizing their effects and preventing them from working properly.

People 18 year of age and older who are participating in a current NEI protocol and meet the following criteria may be eligible for this study:

* Are receiving injections of bevacizumab or ranibizumab for bleeding or swelling in the retina, but the treatment is becoming less effective
* Are receiving injections of bevacizumab or ranibizumab for bleeding or swelling in the retina and the treatment is still effective
* Have bleeding or swelling in the retina, but have never received either bevacizumab or ranibizumab

Participants have blood samples drawn once when they start the study, once in the middle of the study, and once at the end of the study. They are asked permission for study researchers to review the results of their eye examinations at NIH.

DETAILED DESCRIPTION:
Objective

Over the past two years, the field of ophthalmology has witnessed a dramatic paradigm shift in the treatment of exudative and hemorrhagic diseases affecting the retina. This has been due largely to the introduction of two agents, bevacizumab and ranibizumab, into the clinical setting. These agents are humanized monoclonal antibodies which target vascular endothelial growth factor (VEGF). We have observed that, in some patients, a diminished response to these agents occurs with time. One possible explanation for this is the emergence of neutralizing antibodies in patients who have become refractory to bevacizumab or ranibizumab.

Study Population

We will recruit patients from the National Eye Institute (NEI) who are currently receiving treatment with bevacizumab or ranibizumab for various exudative or hemorrhagic disease of the retina. We will also recruit patients with recently diagnosed exudative or hemorrhagic disease of the retina who are na ve to these medications and are going to be treated with them.

Design

This will be a prospective, observational study.

Outcome Measures

The main outcome measure will be the titer of neutralizing antibodies which is measured in patient sera using enzyme-linked immunosorbent assay (ELISA). This will be compared between three groups of patients: 1) 10 patients treated with long term (greater than 1 year) bevacizumab and/or ranibizumab in which decreased drug efficacy has been documented; 2) 10 patients treated with long term (greater than one year) bevacizumab and/or ranibizumab in which decreased drug efficacy has not been documented; and 3) 10 patients who are na ve to treatment with bevacizumab and ranibizumab.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Subjects will include adults being treated for exudative AMD, or macular edema secondary to DR or venous occlusion. The 3 clinical categories, which will each be composed of 10 subjects, are:

  1. Category 1: Patients treated with long term (greater than 1 year) with bevacizumab or ranibizumab in which decreased drug efficacy has been documented. They must have received at least one treatment in the prior 3 months.

     Decreased drug efficacy will be defined as follows: Presence of a therapeutic response (reduction in macula fluid as determined by optical coherence tomography (OCT) or reduction in extent of leakage on fluorescein angiography (FA)) in the first 3 injections, followed by a subsequent decrease in response as evidenced by persistence of intraretinal cysts and/or subretinal fluid on OCT and/or leakage on fluorescein angiography (FA).
  2. Category 2: Patients treated with long term (greater than 1 year) bevacizumab or ranibizumab in which decreased drug efficacy has not been documented. They must have received at least one treatment in the prior 3 months.

     The presence of continued drug efficacy will be defined as follows: Patients who are being treated with bevacizumab or ranibizumab and are demonstrating a good clinical response as demonstrated by the presence of a fluid-free macula on OCT and/or the absence of leakage on FA after treatment.
  3. Category 3: Patients who are na ve to treatment with bevacizumab and ranibizumab

When possible, patients in the 3 categories will be matched by underlying retinal disease type, race, gender, and age.

EXCLUSION CRITERIA:

Patients in the following categories will be excluded from participating in this study:

1. Patients who are currently receiving any form of systemic immunosuppressive or immunomodulatory therapy, including corticosteroids. Immunosuppressive medication could lower the titers of neutralizing that are present in a given patient, and this could give the false impression that such a patient has little to no immune response against bevacizumab or ranibizumab.
2. Patients who have autoimmune or rheumatologic disease. Patients with autoimmune diseases tend to have various autoantibodies in their serum. These naturally present autoantibodies in this patient group could cross-react with bevacizumab or ranibizumab. This would give the false impression that these patients have developed neutralizing antibodies against bevacizumab or ranibizumab, when in fact these naturally occurring cross-reactive autoantibodies were present in the patient all along and are not related to bevacizumab or ranibizumab exposure.
3. Patients with evidence of active systemic infection. Patients with active systemic infection could have various antibodies in the serum, and some of these could cross-react with bevacizumab or ranibizumab. This would give the false impression that these patients have developed neutralizing antibodies against bevacizumab or ranibizumab, when in fact these cross-reactive antibodies were present in the patient secondary to the presence of active systemic infection and are not related to bevacizumab or ranibizumab.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Start 2008-01-16; Primary Completion 2009-08-04 (Actual); Study Completion 2009-08-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Bhisitkul RB. Vascular endothelial growth factor biology: clinical implications for ocular treatments. Br J Ophthalmol. 2006 Dec;90(12):1542-7. doi: 10.1136/bjo.2006.098426. PMID 17114590
- [Background] Noma H, Funatsu H, Yamasaki M, Tsukamoto H, Mimura T, Sone T, Hirayama T, Tamura H, Yamashita H, Minamoto A, Mishima HK. Aqueous humour levels of cytokines are correlated to vitreous levels and severity of macular oedema in branch retinal vein occlusion. Eye (Lond). 2008 Jan;22(1):42-8. doi: 10.1038/sj.eye.6702498. Epub 2006 Jul 7. PMID 16826241
- [Background] Boyd SR, Zachary I, Chakravarthy U, Allen GJ, Wisdom GB, Cree IA, Martin JF, Hykin PG. Correlation of increased vascular endothelial growth factor with neovascularization and permeability in ischemic central vein occlusion. Arch Ophthalmol. 2002 Dec;120(12):1644-50. doi: 10.1001/archopht.120.12.1644. PMID 12470137